CLINICAL TRIAL: NCT06151340
Title: Delayed Language Development in Children With Cleft Palate at Sohag University Hospital
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hadeel Ezeldin Mohamed, Resident Doctor, Sohag University
Other Study IDs: Soh-Med-23-11-06MS
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Delayed Language in Cleft Palate
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — Data collection

SUMMARY:
This is a retrospective study on children with cleft palate who came to the multidisciplinary cleft clinic at Sohag University Hospital from September 2017 to September 2023

ELIGIBILITY:
Inclusion Criteria:

* cleft palate children's

Exclusion Criteria:

* cleft lip only

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: cleft palate children
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Correlation analysis between IQ with degree of delayed language in children with cleft palate (CCP). | 6 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hadeel Ezeldin Mohamed, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No